CLINICAL TRIAL: NCT00871182
Title: A Randomized, Double-blind, Single Dose, Four-period, Six-treatment, Placebo-controlled, Balanced, Incomplete Block, Cross-over, Study of Four Doses of Inhaled PT001 in Patients With Mild to Moderate COPD, Compared to Open Label Tiotropium
Brief Title: Study to Evaluate the Safety and Efficacy of Inhaled PT001 in Patients With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pearl Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PT0010801
Record Dates: First submitted 2009-03-26; First posted 2009-03-30 (Estimated); Last update posted 2013-06-21 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD; obstructive lung diseases; Tiotropium
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive | interventions — Tiotropium Bromide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- PT001 18 mcg (Experimental): Inhaled PT001 18 mcg
  Interventions: Drug: Inhaled PT001
- PT001 36 mcg (Experimental): Inhaled PT001 36 mcg
  Interventions: Drug: Inhaled PT001
- PT001 72 mcg (Experimental): Inhaled PT001 72 mcg
  Interventions: Drug: Inhaled PT001
- PT001 144 mcg (Experimental): Inhaled PT001 144 mcg
  Interventions: Drug: Inhaled PT001
- Inhaled Placebo (Placebo Comparator): Inhaled Placebo
  Interventions: Drug: Inhaled Placebo
- Tiotropium Handihaler (Active Comparator): Tiotropium 18 mcg administered via Handihaler
  Interventions: Drug: Tiotropium Handihaler

INTERVENTIONS:
Drug: Inhaled PT001 — single dose, inhaled
  Arms: PT001 144 mcg; PT001 18 mcg; PT001 36 mcg; PT001 72 mcg
Drug: Inhaled Placebo — single dose, inhaled
  Arms: Inhaled Placebo
Drug: Tiotropium Handihaler — single dose, tiotropium 18 mcg administered via the Handihaler
  Other Names: Spiriva
  Arms: Tiotropium Handihaler

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of inhaled PT001 compared to placebo and tiotropium in patients with mild to moderate chronic obstructive pulmonary disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent
* 40 - 75 years of age
* Females of non-child bearing potential or females of child bearing potential with negative pregnancy test; and acceptable contraceptive methods
* COPD diagnosis
* Current/former smokers with at least a 10 pack-year history of cigarette smoking
* Patients with established clinical history of COPD and severity defined as a post-ipratropium FEV1/FVC ratio of ≤0.70 and FEV1 ≥50 and ≤85% of predicted normal at Screening
* Must demonstrate reversibility to ipratropium demonstrated by a >200 mL improvement over baseline and/or >12% and >150 mL improvement over baseline
* Patients willing to stay at study site for at least 24 hours on each test day

Exclusion Criteria:

* Women who are pregnant or lactating
* Primary diagnosis of asthma
* Alpha-1 antitrypsin deficiency as the cause of COPD
* Active pulmonary diseases
* Prior lung volume reduction surgery
* Abnormal chest X-ray (or CT scan) not due to the presence of COPD
* Hospitalized due to poorly controlled COPD within 24 weeks of Screening
* Unable to perform acceptable spirometry
* Poorly controlled COPD in prior 6-weeks, defined as the occurrence of acute worsening of COPD requiring corticosteroids or antibiotics or acute worsening of COPD requiring treatment prescribed by a physician
* Clinically significant medical conditions
* Symptomatic prostatic hypertrophy or bladder neck obstruction
* Known narrow-angle glaucoma
* Lower respiratory tract infection requiring antibiotics in past 6 weeks
* Clinically significant abnormal ECG
* Clinically significant uncontrolled hypertension
* Positive Hepatitis B surface antigen or Hepatitis C antibody
* Cancer that has not been in complete remission for at least 5 years
* History of hypersensitivity to any beta2-agonists or anticholinergics
* History of severe milk protein allergy
* Known or suspected history of alcohol or drug abuse
* Medically unable to withhold short acting bronchodilators for 6-hours
* Use of the medications below in specified time interval prior to Screening: 3 months: depot corticosteroids, intra-articular corticosteroids; 6 weeks: oral corticosteroids, antibiotics administered for a COPD exacerbation; and 1 month: P-glycoprotein inhibitors, CYP450 3A4 inhibitors, ICS >1000 μg/day of fluticasone propionate or equivalent
* The following COPD medications need to be stopped and switched to appropriate replacement therapies: tiotropium, oral beta2 agonists, LABAs, combination corticosteroid/LABAs, theophylline, leukotriene inhibitors,cromoglycate and nedocromil
* Use of the following medications is prohibited: tricyclic antidepressants, monoamine oxidase (MAO) inhibitors, beta-adrenergic antagonists, anticonvulsants (barbiturates, hydantoins, and carbamazepine and phenothiazines
* Receiving long-term-oxygen or nocturnal oxygen therapy for >12 hours a day
* Diagnosis of sleep apnea that is uncontrolled
* Participation in acute phase of pulmonary rehabilitation in prior 4 weeks
* Will enter acute phase of pulmonary rehabilitation program during study
* Unable to comply with study procedures
* Affiliated with Investigator site
* Questionable validity of consent
* Use of investigational study drug/participation in clinical study in the last 30 days or 5 half lives prior to Screening, whichever is longer

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-03; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Peak improvement in forced expiratory volume in one second (FEV1) | Day 1
  Day 1 serial FEV1 measured over 24 hours

SECONDARY OUTCOMES:
Time to onset of action (>10% improvement in FEV1 from baseline) | Day 1
  Day 1 serial FEV1 measured over 24 hours
Time to peak FEV1 | Day 1
  Day 1 serial FEV1 measured over 24 hours
FEV1 area under the curve (AUC) from 0 to 24 hours | Day 1
  Day 1 serial FEV1 measured over 24 hours
FEV1 AUC from 0 to 12 hours | Day 1
  Day 1 serial FEV1 measured over 24 hours
Trough FEV1 at 12 and 24 hours | Day 1
  Day 1 serial FEV1 measured over 24 hours
Peak Improvement in inspiratory capacity (IC) | Day 1
  Day 1 serial IC measured over 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Colin Reisner, M.D., Study Director — Pearl Therapeutics, Inc.
Locations (6):
- United States (6):
  - Pivotal Research Centers, Peoria, Arizona
  - National Jewish Health, Denver, Colorado
  - Elite Research Institute, Miami, Florida
  - Pulmonary and Critical Care Medicine, Omaha, Nebraska
  - Cincinnati VAMC, Cincinnati, Ohio
  - Spartanburg Medical Research, Spartanburg, South Carolina

REFERENCES:
- [Derived] Rennard S, Fogarty C, Reisner C, Fernandez C, Fischer T, Golden M, Rose ES, Darken P, Tardie G, Orevillo C. Randomized study of the safety, pharmacokinetics, and bronchodilatory efficacy of a proprietary glycopyrronium metered-dose inhaler in study patients with chronic obstructive pulmonary disease. BMC Pulm Med. 2014 Jul 16;14:118. doi: 10.1186/1471-2466-14-118. PMID 25027304